CLINICAL TRIAL: NCT05353543
Title: Acupuncture Therapy Based on Biological Specificity of Acupoints for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: The Zhejiang Provincial Tongde Hospital (Unknown); The Affiliated Hangzhou First People's Hospital (Unknown)
Responsible Party: Principal Investigator, Xiaomei Shao, Prof, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-ABS
Record Dates: First submitted 2022-04-27; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder
Keywords: acupuncture; biological specificity; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (strong reaction acupoints) group (Experimental): This group will include 40 patients with MDD who will be treated with acupuncture and SSRIs antidepressants. Strong reaction acupoints selected in the first part of the study will be stimulated. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Drug: SSRIs; Procedure: acupuncture (strong reaction acupoints)
- Acupuncture (weak reaction acupoints) group (Experimental): This group will include 40 patients with MDD who will be treated with acupuncture and SSRIs antidepressants. Weak reaction acupoints selected in the first part of the study will be stimulated. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Drug: SSRIs; Procedure: acupuncture (weak reaction acupoints)
- Sham acupuncture group (Experimental): This group will include 40 patients with MDD who will be treated with sham acupuncture and SSRIs antidepressants. The sham acupuncture will be needled on the points 1cm lateral to strong reaction acupoints. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Drug: SSRIs; Procedure: sham acupuncture

INTERVENTIONS:
Drug: SSRIs — In this study, SSRIs antidepressants will be used, and the oral dose will be determined by the clinical specialist. Once-daily for 6 weeks.
  Other Names: SSRIs antidepressants
Procedure: acupuncture (strong reaction acupoints) — This study will use the intradermal needle as an acupuncture intervention. Strong reaction acupoints selected in the first part of the study will be stimulated. According to the position of the acupoints, choose a needle of φ0.20*1.5m or φ0.20*1.2mm. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: intradermal needle
  Arms: Acupuncture (strong reaction acupoints) group
Procedure: acupuncture (weak reaction acupoints) — This study will use the intradermal needle as an acupuncture intervention. Weak reaction acupoints selected in the first part of the study will be stimulated. According to the position of the acupoints, choose a needle of φ0.20*1.5m or φ0.20*1.2mm. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: intradermal needle
  Arms: Acupuncture (weak reaction acupoints) group
Procedure: sham acupuncture — Sham acupuncture will use the same size, color, and material as the verum intradermal needle with a thin silicone pad in the middle instead of the needle body. The sham acupuncture will be needled on the points 1cm lateral to strong reaction acupoints. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. A total of 10 sessions will be performed for 6 weeks.
  Other Names: sham intradermal needle
  Arms: Sham acupuncture group

SUMMARY:
Acupoints are the stimulus points and reactive points for acupuncture to treat the diseases. Therefore, this study is designed to detect the biological specificity of acupoints in healthy participants and major depressive disorder (MDD) participants by using multiple objective assessment tools. And then acupoints that are statistically different between the two groups will be defined as strong reaction points, and other acupoints without statistically different will be defined as weak response points. In addition, this clinical trial will be conducted to explore whether the efficacy of stimulating strong reaction acupoints is more effective than weak reaction points, thereby confirming the specificity of the acupoint.

DETAILED DESCRIPTION:
Part 1: This study will include 40 patients with MDD and 40 healthy control participants. Infrared thermography (IRT), laser doppler flowmetry (LDF), functional near-infrared spectroscopy (FNIS), and digital pressure pain gauge (PPG), respectively, will be adopted to assess 4 kinds of biological specificity of MDD related acupoints, namely, the thermal transport specificity, the microcirculatory specificity, the metabolic specificity, and the pain sensitivity specificity. Based on the results of this study, we will select acupoints with statistical differences between the two groups as the strong reaction acupoints and the remaining acupoints as the weak reaction acupoints.

Part 2: A total of 120 participants with MDD who meet the inclusion criteria will be included in the study. All participants will receive basic treatment of selective serotonin reuptake inhibitors (SSRIs) antidepressants. They will be randomly divided into the acupuncture (strong reaction acupoints) group, acupuncture (weak reaction acupoints) group, and sham acupuncture group. We will evaluate the therapeutic effect and safety of acupuncture for MDD, furthermore, to demonstrate whether stimulating strong reaction acupoints has more advantages in the treatment of MDD than weak reaction acupoints.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for health volunteers:

   * Healthy volunteers who could provide a recent depression screening report, and confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine, or neurological disease;
   * 12 ≤ age ≤60 years, male or female;
   * Participants have clear consciousness and could communicate with others normally;
   * Participants could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin (for minor participants, their guardian should sign the informed consent form for them).
2. Inclusion criteria for MDD:

   * Patients should meet the diagnostic criteria of the International Classification of Diseases 10th Edition (ICD-10) diagnostic criteria for depression and are evaluated as moderate or severe MDD according to the severity of depression;
   * 12 ≤ age ≤60, male or female;
   * Participants have clear consciousness and could communicate with others normally;
   * Participants could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin (for minor participants, their guardian should sign the informed consent form for them).

Exclusion Criteria:

1. Exclusion criteria of health volunteers:

   * Participants with serious primary diseases of cardiovascular diseases, liver diseases, kidney diseases, urinary diseases, and hematological diseases;
   * Participants have a mental illness, alcohol dependence, or a history of drug abuse;
   * Pregnant or lactating participants;
   * Participants are participating in other trials.
2. Exclusion criteria for MDD:

   * Participants with serious primary diseases of cardiovascular, respiratory, digestive, urinary, hematological, endocrine, neurological disease, and other serious primary diseases, and the disease cannot be effectively controlled clinically;
   * Major depressive disorders caused by organic mental disorders, schizophrenia, bipolar disorder, psychoactive substances, and non-addictive substances;
   * Participants with suicidal tendencies;
   * Pregnant or lactating participants;
   * Participants taking other antidepressants that were not SSRIs or the pharmacological effects of such antidepressants have not been cleared;
   * Participants with intellectual disabilities who cannot cooperate with the questionnaire survey;
   * Participants with bleeding tendency, skin disease, allergic constitution, and allergic to adhesive tape;
   * The skin at the test site of participants has scars, hyperpigmentation, red and swollen;
   * Participants are participating in other trials.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionaire-9 Items (PHQ -9) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The PHQ-9 scale has a total of 9 questions, each with a score of 0-3 (none: 0; a few days: 1; more than half of the time: 2; almost every day: 3), with a total score of 0-27.

SECONDARY OUTCOMES:
Change in the Self-Rating Depression Scale (SDS) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  This scale has 20 questions. Participants should choose the answer that best matches their situation based on their feelings in the last week or less. Depression severity = total score/80 (0-0.5 means no depression, 0.5-0.59 means mild depression, 0.6-0.69 means moderate depression, and 0.7 or more means severe depression).
Temperature change | Baseline, 6 weeks after treatment.
  NEC R450 Infrared thermography will be used to record baseline temperature and the temperature change of relevant sites. The average temperature value of relevant sites in the six infrared thermograms is its base temperature.
Microcirculatory change | Baseline, 6 weeks after treatment.
  The PeriFlux System 5000 is a four-channel laser Doppler flowmeter that detects the rate of blood cell movement and its distribution of relevant test sites. The accompanying Perisoft for Windows flow analysis software generates the blood flow curve and analyzes the microcirculatory perfusion unit (PU) at the relevant test site and the 10 min average is used as the base PU.
Metabolic change | Baseline, 6 weeks after treatment.
  The INVOS 5100C quad-channel NIR spectrometer detects regional oxygen saturation (rSO2). rSO2 is analyzed by the INVOS Analytics Tool software and the 10 min average is used as the base rSO2.
Pain sensitivity change | Baseline, 6 weeks after treatment.
  A Digital pressure pain gauge will be used to measure the local pain threshold (PT). The probe of the pain gauge will be placed vertically on the relevant test site, and the pressure will be applied slowly and steadily, and when the participant feels pain, the pressure will stop and the reading on the gauge is the PT. The average value of the PT of the same relevant test sites will be calculated as their base PT.
Adverse Events | Up to 10 weeks
  Any adverse events that occur during the trial will be recorded and analyzed for the cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No